CLINICAL TRIAL: NCT05578586
Title: A Pilot Study for Optimizing Meropenem Administration in the Intensive Care Unit - Short Six Times vs Prolonged Three Times Courses Daily
Brief Title: A Pilot Study for Optimizing Meropenem Administration in the ICU
Acronym: MER6
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ingvild Nordøy, Senior consultant, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meropenem6
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Drug Effect
MeSH Terms: interventions — Meropenem

STUDY DESIGN:
Intervention Model Description: Prospective randomized pilotstudy 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental vs Control (Experimental): The patients who are randomized to receive meropenem 1 gram 6 times daily in 15 minutes infusions.
  Interventions: Drug: Meropenem 1000 mg
- Controls (Active Comparator): The patients who are randomized to receive meropenem 2 gram 3 times daily in 3 hours infusions.
  Interventions: Drug: Meropenem 1000 mg

INTERVENTIONS:
Drug: Meropenem 1000 mg — given as 6 or 3 infusions in 15 minues or 3 hours.
  Other Names: Meropenem 2000 mg

SUMMARY:
Can antibiotic drugs be administered faster and make acceptable serum concentrations if we give short but multiple infusions compared to long and fewer infusions? In this study we will compare giving meropenem 1 gram 6 times daily in 15 minutes infusions to the recommended 2 gram 3 times daily in 3 hours infusions. In patients in the intensive care unit, the need for intravenous access is of essence. If 6 short infusions results in the same serum concentrations as 3 long infusions, we will increase intravenous access from 15 to 22.5 hours daily.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to examine if the dosing of the antibiotic meropenem given as 1 gram 6 times daily in 15 minutes infusions can be compared to 2 grams given 3 times daily in 3 hours infusion when measuring the serum concentration above the minimum inhibitory concentration (MIC) ≥ 50 % of the time (2 mg/l).

The secondary aims are

* That both administration forms will result in serum concentrations above MIC ≥ 100 % of the time (2 mg/l)
* Days in hospital
* 30 days mortality after admittance to the ICU
* Serious side-effects

Five extra blood samples will be performed 24, 48 and 72 hours between two dosing intervals. The dose will be adjusted according to renal function which will be monitored daily. The patients will be supervised for adverse effects until 2 days after treatment has stopped.

The study will be performed from 2021 to the end of 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years admitted to the ICU at Oslo University Hospital, Rikshospitalet and
2. who shall be treated with meropenem because of proven or suspected serious infection and
3. who give their written informed consent either directly or through next of kin

Exclusion Criteria: Patients

1. with known hypersensistivity to betalactam antibiotics or
2. who use of valproat or
3. who are pregnant or
4. the lack of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Concentration above the minimum inhibitory concentration (MIC) ≥ 50 % of the time (2 mg/l) | After 24, 48 and 72 hours
  Comparing 2 ways of administering meropenem intravenously

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild Nordøy, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turnidge JD. The pharmacodynamics of beta-lactams. Clin Infect Dis. 1998 Jul;27(1):10-22. doi: 10.1086/514622. PMID 9675443
- [Result] Craig WA. Pharmacokinetic/pharmacodynamic parameters: rationale for antibacterial dosing of mice and men. Clin Infect Dis. 1998 Jan;26(1):1-10; quiz 11-2. doi: 10.1086/516284. PMID 9455502
- [Result] Drusano GL. Antimicrobial pharmacodynamics: critical interactions of 'bug and drug'. Nat Rev Microbiol. 2004 Apr;2(4):289-300. doi: 10.1038/nrmicro862. No abstract available. PMID 15031728
- [Result] Roberts JA, Lipman J. Optimizing use of beta-lactam antibiotics in the critically ill. Semin Respir Crit Care Med. 2007 Dec;28(6):579-85. doi: 10.1055/s-2007-996404. PMID 18095221
- [Result] De Waele JJ, Lipman J, Carlier M, Roberts JA. Subtleties in practical application of prolonged infusion of beta-lactam antibiotics. Int J Antimicrob Agents. 2015 May;45(5):461-3. doi: 10.1016/j.ijantimicag.2015.01.007. Epub 2015 Feb 16. PMID 25749200
- [Result] Roberts JA, Paul SK, Akova M, Bassetti M, De Waele JJ, Dimopoulos G, Kaukonen KM, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Starr T, Wallis SC, Lipman J; DALI Study. DALI: defining antibiotic levels in intensive care unit patients: are current beta-lactam antibiotic doses sufficient for critically ill patients? Clin Infect Dis. 2014 Apr;58(8):1072-83. doi: 10.1093/cid/ciu027. Epub 2014 Jan 14. PMID 24429437
- [Result] Taccone FS, Laterre PF, Dugernier T, Spapen H, Delattre I, Wittebole X, De Backer D, Layeux B, Wallemacq P, Vincent JL, Jacobs F. Insufficient beta-lactam concentrations in the early phase of severe sepsis and septic shock. Crit Care. 2010;14(4):R126. doi: 10.1186/cc9091. Epub 2010 Jul 1. PMID 20594297
- [Result] Binder L, Schworer H, Hoppe S, Streit F, Neumann S, Beckmann A, Wachter R, Oellerich M, Walson PD. Pharmacokinetics of meropenem in critically ill patients with severe infections. Ther Drug Monit. 2013 Feb;35(1):63-70. doi: 10.1097/FTD.0b013e31827d496c. PMID 23318279
- [Result] Petersson J, Giske CG, Eliasson E. Standard dosing of piperacillin and meropenem fail to achieve adequate plasma concentrations in ICU patients. Acta Anaesthesiol Scand. 2016 Nov;60(10):1425-1436. doi: 10.1111/aas.12808. Epub 2016 Sep 21. PMID 27655029
- [Result] Mouton JW, Ambrose PG, Canton R, Drusano GL, Harbarth S, MacGowan A, Theuretzbacher U, Turnidge J. Conserving antibiotics for the future: new ways to use old and new drugs from a pharmacokinetic and pharmacodynamic perspective. Drug Resist Updat. 2011 Apr;14(2):107-17. doi: 10.1016/j.drup.2011.02.005. Epub 2011 Mar 26. PMID 21440486
- [Result] Roberts JA, Abdul-Aziz MH, Davis JS, Dulhunty JM, Cotta MO, Myburgh J, Bellomo R, Lipman J. Continuous versus Intermittent beta-Lactam Infusion in Severe Sepsis. A Meta-analysis of Individual Patient Data from Randomized Trials. Am J Respir Crit Care Med. 2016 Sep 15;194(6):681-91. doi: 10.1164/rccm.201601-0024OC. PMID 26974879
- [Result] Roberts JA, Webb S, Paterson D, Ho KM, Lipman J. A systematic review on clinical benefits of continuous administration of beta-lactam antibiotics. Crit Care Med. 2009 Jun;37(6):2071-8. doi: 10.1097/CCM.0b013e3181a0054d. PMID 19384201
- [Result] Falagas ME, Tansarli GS, Ikawa K, Vardakas KZ. Clinical outcomes with extended or continuous versus short-term intravenous infusion of carbapenems and piperacillin/tazobactam: a systematic review and meta-analysis. Clin Infect Dis. 2013 Jan;56(2):272-82. doi: 10.1093/cid/cis857. Epub 2012 Oct 16. PMID 23074314
- [Result] Teo J, Liew Y, Lee W, Kwa AL. Prolonged infusion versus intermittent boluses of beta-lactam antibiotics for treatment of acute infections: a meta-analysis. Int J Antimicrob Agents. 2014 May;43(5):403-11. doi: 10.1016/j.ijantimicag.2014.01.027. Epub 2014 Mar 1. PMID 24657044
- [Result] Ahmed N, Jen SP, Altshuler D, Papadopoulos J, Pham VP, Dubrovskaya Y. Evaluation of Meropenem Extended Versus Intermittent Infusion Dosing Protocol in Critically Ill Patients. J Intensive Care Med. 2020 Aug;35(8):763-771. doi: 10.1177/0885066618784264. Epub 2018 Jun 28. PMID 29954243